CLINICAL TRIAL: NCT02994498
Title: An Open-Label Phase I/IIa Dose-Escalation Study Evaluating the Safety, Tolerability and Efficacy of DCB-BO1301 as Add-on Therapy to Dacarbazine in Subjects With Advanced Melanoma
Brief Title: Safety and Efficacy of DCB-BO1301 in Advanced Melanoma
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chung Mei Biopharma Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CMB-B01
Record Dates: First submitted 2016-12-09; First posted 2016-12-16 (Estimated); Last update posted 2022-03-18 (Actual); Status verified 2022-03

CONDITIONS: Advanced Melanoma

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- DCB-BO1301 1 capsule (Experimental): DCB-BO1301 1 capsule, tid (around 1 hour before meal) for at most 48 weeks
  Interventions: Drug: DCB-BO1301
- DCB-BO1301 2 capsules (Experimental): DCB-BO1301 2 capsules, tid (around 1 hour before meal) for at most 48 weeks
  Interventions: Drug: DCB-BO1301
- DCB-BO1301 3 capsules (Experimental): DCB-BO1301 3 capsules, tid (around 1 hour before meal) for at most 48 weeks
  Interventions: Drug: DCB-BO1301

INTERVENTIONS:
Drug: DCB-BO1301 — 1, 2, or 3 capsules, three times a day, oral, at most 48 weeks

SUMMARY:
The primary study objectives are

1. to evaluate the safety and tolerability profiles of DCB-BO1301 and to determine the maximum tolerated dose (MTD) of DCB-BO1301 as add-on therapy to dacarbazine in subjects with advanced melanoma (Phase I)
2. to evaluate the efficacy profile of DCB-BO1301 at MTD or lower dose level as add-on therapy to dacarbazine in subjects with advanced melanoma in terms of progression free survival (Phase IIa)

ELIGIBILITY:
Inclusion Criteria:

1. Subjects ≧ 20 years old (inclusive)
2. Histologically or cytologically confirmed advanced melanoma, (stage III or IV)
3. Subject must have at least one of the following:

   * Melanoma that was previously treated with at least one complete or partial course of therapy for melanoma with either a poor to no response or evidence of disease progression;
   * Melanoma that cannot be treated with first-line therapies because of medical comorbidities/risk of toxicity; or
   * Melanoma that has not been treated with first-line therapies because of patient refusal.
4. If melanoma is possibly resectable, the melanoma must have recurred despite at least two attempts at resection.
5. Evaluable disease, at least one measurable target lesion on imaging by RECIST 1.1 criteria on previous scan
6. ECOG performance status ≤ 2 and life expectancy ≥ 3 months Note: ECOG = Eastern Cooperative Oncology Group
7. Females subjects must be either

   * of non-childbearing potential:
   * Or, if of childbearing potential:

     * Must have a negative urine or serum pregnancy test at screening, and
     * If heterosexually active, must use at least 1 form of birth control (which must be a barrier method) starting at screening and through the primary study period.
8. Female subject must not be breastfeeding at screening, through the treatment period and through the primary study period.
9. Male subject and their female spouse/partners who are of childbearing potential must be using highly effective contraception consisting of 2 forms of birth control (1 of which must be a barrier method) starting at screening, through the treatment period and through the primary study period.
10. Dated and signed informed consent

Exclusion Criteria:

1. Primary CNS malignancies or clinically active CNS metastases
2. Ascertained hypersensitivity to any component of investigational product or standard therapies that the subject will be treated
3. Any of the following hematologic abnormalities:

   1. Hemoglobin < 10 g/dL,
   2. ANC < 1,500/μL,
   3. Platelets < 75,000 /μL Note: ANC = absolute neutrophil count
4. Any of the following serum chemistry abnormalities:

   1. Total bilirubin > 1.5 × ULN,
   2. AST, ALT, or Alk-P > 2.5 × ULN,
   3. serum albumin < 2.5 g/dL,
   4. creatinine > 1.5 × ULN,
   5. creatine phosphokinase (CPK) > 2.5 × ULN,

   d. any other ≥ Grade 3 laboratory abnormality at baseline (other than those listed above) Note: ULN = upper limit of normal. AST = aspartate transaminase, ALT = alanine transaminase
5. History of known brain metastases
6. Anticipated requiring, being taking, or taken with past 2 weeks of Screening visit of systemic steroid, immunosuppressive agents, aspirin (more than 100 mg/day), NSAID (except COX-2 Inhibitors), heparin, low molecular weight heparin or warfarin (more than 1 mg/day) Note: NSAID = Nonsteroidal anti-inflammatory drugs
7. Uncontrolled nausea or vomiting or any symptom that would prevent the ability to comply with daily oral DCB-BO1301 treatment
8. Serious/active infection such as HIV, HBV or HCV carrier, or infection requiring parenteral antibiotics Note: HIV = Human immunodeficiency virus; HBV = Hepatitis B virus; HCV = hepatitis C virus
9. Uncontrolled psychiatric disorder or altered mental status precluding informed consent or necessary testing
10. Consumption of herbal preparations/supplements (except for a daily multivitamin/mineral supplement not containing herbal components) within 2 weeks prior to the start of DCB-BO1301 administration
11. Significant cardiovascular disease, including:

    1. Active clinically symptomatic left ventricular failure
    2. Active hypertension (diastolic blood pressure > 100 mmHg). Subjects with a history of hypertension must have been on stable doses of anti-hypertensive drugs for ≥ 4 weeks prior to start of DCB-BO1301 administration
    3. Uncontrolled hypertension: Blood pressure >140/90 mmHg on more than 2 antihypertensive medications
    4. Myocardial infarction within 3 months prior to the start of DCB-BO1301 administration
    5. Prothrombin time > 1.5 x ULN; APTT abnormal (< 20 sec or > 34 sec) ; long QT syndrome
12. Significant gastrointestinal disorder(s) that would, in the opinion of the investigator, prevent absorption of an orally available agent
13. Has received an investigational agent within 4 weeks of entering this study
14. With any condition judged by the investigator that entering the trial may be detrimental to the subject
15. Receiving chemotherapy, investigational or hormonal therapy, major surgeries in the previous 4 weeks of Screening visit.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2023-03 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose | Week 6

SECONDARY OUTCOMES:
Incidence of adverse events | Weeks 3, 6, 9, 12, 15, 18, 21, 24, 27, 30, 33, 36, 39, 42, 45, 48, 52
Response rate | Weeks 3, 6, 9, 12, 15, 18, 21, 24, 27, 30, 33, 36, 39, 42, 45, 48, 52
Overall survival | Weeks 3, 6, 9, 12, 15, 18, 21, 24, 27, 30, 33, 36, 39, 42, 45, 48, 52, 64, 76
Changes in global health/QoL standardized score at post-treatment visits compared to baseline. | Weeks 0, 3, 6, 9, 12, 15, 18, 21, 24, 27, 30, 33, 36, 39, 42, 45, 48, 52
Progression free survival | Weeks 0, 3, 6, 9, 12, 15, 18, 21, 24, 27, 30, 33, 36, 39, 42, 45, 48, 52, 64,76